CLINICAL TRIAL: NCT00489034
Title: Drug Use and HIV-Infected Female Adolescents' Care Use
Brief Title: Engaging Care for HIV-infected Adolescent Females.
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 009; 1R01DA014706-01 (NIH)
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-08

CONDITIONS: HIV Infection
Keywords: HIV; adolescent females; adherence; clinical care; risk behaviors
MeSH Terms: conditions — HIV Infections; Risk-Taking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Index Participants: HIV-infected females, ages 13- 23 years, recruited from ATN sites in New York, Chicago, Miami, Los Angeles, and New Orleans will undergo quantitative interviewing. A sub-sample of the group will undergo ethnographic and/or gender interviewing.
  Interventions: Behavioral: Quantitative Interview; Behavioral: Ethnographic Interview; Behavioral: Gender Interview
- Network Participants: Closest friends of index participants s and parents/guardians of index participants who know the index participant's HIV status will undergo quantitative interviewing. A sub-sample of the group will undergo ethnographic interviewing.
  Interventions: Behavioral: Quantitative Interview; Behavioral: Ethnographic Interview

INTERVENTIONS:
Behavioral: Quantitative Interview — Index participants will be interviewed every six months (with phone interviews focused on service utilization at each six month interval midpoint) for 18 months while network members will be interviewed at baseline and one year. Interviews will consist of in-depth face-to-face and audio computer-assisted interviews (ACASIs) and a structured diagnostic interview to assess engagement in care (number of clinical visits attended), substance use, attitudes about substance use, friend's substance use, sexual risk behaviors, PTSD (for index participants only), support of index participants care use (network participants only), attitudes about healthcare (network participants only), index participant's adherence (network participants only), own functioning (network participants only), and family functioning (network participants only). At Baseline only, a urine sample will be collected from index participants for drug testing to assess the agreement between urine and ACASI.
Behavioral: Ethnographic Interview — Qualitative interviews will be conducted with a small sub-sample of index and identified network participants from each site at least monthly for a period of 18 months. Interviews will be ethnographic in nature and will rely on participants' life stories and narratives of social experience to supply their content and guide their progression.
Behavioral: Gender Interview — Qualitative interviews will be conducted with a sub-sample of index participants. These interviews will focus on issues of gender related vulnerabilities and will be used to develop a survey.
  Groups: Index Participants

SUMMARY:
The proposed multi-site, longitudinal study will examine the correlation of substance use, mental health disorders, and social networks to engagement in care for HIV-infected adolescent females, aged 13 years, 0 months - 23 years, 11 months, and suggest ways to promote adherence and retention in treatment, care, and prevention programs. Qualitative and quantitative data collection methods will be used with index participants and network members.

DETAILED DESCRIPTION:
The primary outcome examined in the proposed study is engagement in care, operationalized as the number of clinical visits attended. Clinic visits will be monitored on a weekly basis. Secondary outcomes of interest include medication adherence, sexual risk behaviors, and substance use. For the quantitative study, formal psychological testing will be conducted with index adolescent females, and biological specimens will be collected to validate self-reported drug use. CD-4 counts and viral load will be monitored every three months via chart review.

Index adolescents will be interviewed every six months (with phone interviews focused on service utilization at each six month interval midpoint) for eighteen months while network members will be interviewed at baseline and one year.

Qualitative interviews in the Ethnographic Study will be conducted with a small sub-sample of index and identified network participants from each site at least monthly for a period of at least 18 months. Qualitative interviews will be ethnographic in nature and will rely on participants' life stories and narratives of social experience to supply their content and to guide their progression.

Qualitative Interviews in the Gender Substudy will be conducted with a subsample of index participants. These qualitative interviews will focus on issues of gender related vulnerabilities and will be used to develop a survey to be administered to all index participants from sites participating in this substudy.

ELIGIBILITY:
Quantitative Study Inclusion Criteria

Index Participants:

1. Female.
2. Age 13 years, 0 months - 23 years, 11 months (364 days).
3. All race/ethnicities.
4. English or Spanish speaking.
5. Non-perinatal, non-transfusion acquired HIV.
6. Unknown transmission status with study personnel approval.

Network Participants:

Parents/Guardians of Index Participants:

1. Know patient's HIV status
2. Male or female.
3. All race/ethnicities
4. English or Spanish speaking.
5. Serve a parental or guardian-like role.

Close Friend of Index Participants:

1. Close friend of index subject.
2. Male or female.
3. Minimum age 13 years, 0 months.
4. All race/ethnicities
5. English or Spanish speaking

Ethnographic Sub-Sample

Inclusion Criteria:

Index Participants:

1. Enrolled in Quantitative NIDA study.
2. English-speaking at Miami, New York, Chicago, and New Orleans sites.
3. English or Spanish-speaking at Los Angeles USC site

Network Participants:

1. English-speaking at Miami, New York, Chicago, and New Orleans sites.
2. English or Spanish-speaking at Los Angeles USC site.
3. Know index serostatus.

Gender Sub-Sample

Inclusion Criteria:

1. Age 18 years, 0 months - 23 years, 11 months.
2. Enrolled in quantitative study.
3. English-speaking.
4. Female.

Ages: 13 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-infected adolescent females, aged 13 years, 0 months - 23 years, 11 months will be followed to examine the correlation of substance use, mental health disorders, and social networks to engagement in care and suggested ways to promote adherence and retention in treatment, care, and prevention.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2003-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Engagement in Care among Index Participants | Baseline, 6 months, 12 months, and 18 months
  Engagement in care will be operationalized as the number of clinic visits attended and will be assessed through the qualitative interviews.

SECONDARY OUTCOMES:
Medication Adherence | Baseline, 6 months, 12 months, and 18 months
  As assessed through the qualitative interviews for index and network participants.
Sexual Risk Behaviors | Baseline, 6 months, 12 months, and 18 months
  As assessed through the qualitative interviews for index and network participants.
Substance Use | Baseline, 6 months, 12 months, and 18 months
  As assessed through the qualitative interviews for index and network participants.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Perez, Ph.D, Study Director — Westat
Locations (5):
- United States (5):
  - Universtiy of Southern California, Los Angeles, California
  - University of Miami, School of Medicine, Miami, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Adolescent Medicine Trials Network for HIV/AIDS Interventions Website — http://www.atnonline.org